CLINICAL TRIAL: NCT04258631
Title: Wound Infiltration With Liposomal Bupivacaine With or Without Intrathecal Analgesia in Laparotomy for Gynecological Malignancy: A Randomized Controlled Trial
Brief Title: Liposomal Bupivacaine With or Without Hydromorphone for the Improvement of Pain Control After Laparotomy in Patients With Gynecological Malignancies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MC2061; NCI-2020-00609 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-010500 (Other: Mayo Clinic Institutional Review Board); MC2061 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Malignant Female Reproductive System Neoplasm
MeSH Terms: interventions — Hydromorphone; Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (laparotomy, liposomal bupivacaine) (Active Comparator): Patients undergo standard of care laparotomy and then receive liposomal bupivacaine.
  Interventions: Procedure: Laparotomy; Drug: Liposomal Bupivacaine; Other: Questionnaire Administration
- Arm II (laparotomy, liposomal bupivacaine, hydromorphone) (Experimental): Patients undergo standard of care laparotomy and then receive liposomal bupivacaine and hydromorphone IT.
  Interventions: Drug: Hydromorphone; Procedure: Laparotomy; Drug: Liposomal Bupivacaine; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Hydromorphone — Given IT
  Other Names: (-)-Hydromorphone; Dihydromorphinone; Hydromorphon
  Arms: Arm II (laparotomy, liposomal bupivacaine, hydromorphone)
Procedure: Laparotomy — Undergo laparotomy
Drug: Liposomal Bupivacaine — Drug
  Other Names: Bupivacaine Liposome Injectable Suspension; Exparel
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase IV trial studies how well liposomal bupivacaine with or without hydromorphone works in improving pain control during the first 24 hours after surgery in patients with gynecological malignancies undergoing laparotomy. Liposomal bupivacaine is routinely infiltrated into the skin surrounding the abdominal incision, and is effective in providing good relief of incisional pain. Hydromorphone is also a type of pain medication that may provide better management of deep abdominal pain. It is not yet known if giving liposomal bupivacaine with or without hydromorphone will work better in improving pain in patients with gynecological malignancies during the first 24 hours after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate if no additional intervention is noninferior to intrathecal analgesia (ITA) for postoperative pain experience 24 hours after surgery after laparotomy for gynecological malignancy within an established enhanced recovery pathway which includes incisional liposomal bupivacaine (ILB).

II. Evaluate the effect of intrathecal analgesia on patient satisfaction with postoperative analgesia after laparotomy for gynecological malignancy.

III. Report the impact of ITA use on cost. IV. Validate the Quality of Recovery (QOR)-15 in our population.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo standard of care laparotomy and then receive liposomal bupivacaine.

ARM II: Patients undergo standard of care laparotomy and then receive liposomal bupivacaine and hydromorphone intrathecally (IT).

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery for suspected (based on consulting surgeon's opinion-imaging, laboratory [lab], pathology [path]) gynecological malignancy, enhanced recovery after surgery (ERAS) protocol

Exclusion Criteria:

* Inability to read or understand English
* Prehospitalization narcotic use if weekly average daily oral morphine equivalent of > 20 mg
* Chronic pain syndromes such as fibromyalgia
* Extensive surgery planned (surrogate for post-operative [postop] pain): Planned intensive care unit (ICU) admission, abdominoperineal resection, exenteration, use of intraoperative radiation (IORT), hyperthermic intraperitoneal chemotherapy (HIPEC)
* Contraindication to neuraxial analgesia:

  * Coagulopathy

    * International normalized ratio (INR) > 1.2 current or predicted after surgery (e.g. planned right hepatic resection)
    * Thrombocytopenia. Platelets (plts) < 100
    * Hemophiliac disease states (hemophilia, von Willebrand disease, etc.)
    * Patients receiving antithrombotic or thrombolytic therapy are excluded according to the American Society of Regional Anesthesia and Pain Medicine (ASRA) guidelines
  * Localized infection at the potential site of injection
  * Significant developmental or structural spinal abnormalities that would preclude a safe spinal technique. These include spina bifida, tethered spinal cord, lumbar spinal fusion, and active lumbar radiculopathy
* Patients with stage 4 or 5 kidney disease (glomerular filtration rate [GFR] less than 30 ml/min per 1.73 m^2)
* Intolerance or allergy to opioids, acetaminophen, or amide-type local anesthetics
* Current pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean C Dowdy, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Started | 59 | 46
Completed | 59 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone) | Total
Number analyzed (Participants) | 59 | 46 | 105
Age, Categorical [Count of Participants; unit: Participants] — Age recorded at the time of surgery.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 31 | 24 | 55
    >=65 years | 28 | 22 | 50
Age, Continuous [Median (Full Range); unit: years] | 56 [34 to 78] | 56.5 [37 to 76] | 56 [34 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 46 | 105
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 55 | 46 | 101
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 55 | 46 | 101
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 59 | 46 | 105

OUTCOME MEASURES:

1. Primary Outcome: Overall Benefit of Analgesia Score (OBAS)
Description: The Overall Benefit of Analgesia Score (OBAS) is a multi-dimensional survey that measures a patient's benefit from postoperative pain therapy. It assesses pain intensity, opioid-related adverse events, and patient satisfaction with analgesia. Each of 7 questions are scored on a scale from 0 to 4 where 0=minimal/not at all and 4=maximum/very much. The total score is a sum of the 7 item scores with question 7 scored as 4 minus the patient reported number. Total scores range from 0 to 28 with lower scores representing greater benefit from analgesic therapy. The median total OBAS score for each group is presented.
Time Frame: Up to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
score on a scale | 4 [2 to 7] | 4 [3 to 9]

2. Secondary Outcome: Cumulative 24-hour Narcotic Consumption
Description: Various narcotic medications are standardized and reported as Morphine Milligram Equivalents (MME).
Time Frame: Up to 24 hours after surgery
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
Morphine Milligram Equivalents (MME) | 41.4 (31.9) | 17.5 (25.0)

3. Secondary Outcome: Post-operative Pain Scores
Description: Postoperative pain is scored on a scale of 0 - 10, with the lower score showing a better outcome.
Time Frame: Up to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
score on a scale | 4 [2.5 to 5] | 3 [1 to 5]

4. Secondary Outcome: Time to First Analgesic Request
Description: Amount of time from leaving surgery to the first request for pain relief.
Time Frame: Up to 24 hours after surgery
Population: Analyses were based on treatment received, not randomization arm.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
minutes | 20.1 [2.5 to 35.0] | 25.0 [2.5 to 38.0]

5. Secondary Outcome: Use of Intravenous (IV) Patient-controlled Analgesia
Description: Number of patients that used IV, patient controlled analgesia after surgery.
Time Frame: Up to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
Participants | 3 | 5

6. Secondary Outcome: Use of Intravenous Rescue Opioids
Description: Number of patients that needed IV rescue opioids after surgery.
Time Frame: Up to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
Participants | 42 | 12

7. Secondary Outcome: Length of Stay
Description: Length of associated hospitalization in days.
Time Frame: Up to 1 week after surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
days | 3.8 [2.9 to 4.9] | 3.4 [2.1 to 4.9]

8. Secondary Outcome: Additional Fluid Requirement After 24 Hours of Surgery
Description: Number of patients requiring additional IV fluids after surgery.
Time Frame: Up to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
Participants | 27 | 24

9. Secondary Outcome: Weight Gain Following Surgery
Description: Weight difference post- and pre-surgery.
Time Frame: Up to 24 hours after surgery
Population: Data not collected
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Total Cost of Care
Description: All medical costs occurring during hospitalization.
Time Frame: Entire hospitalization, approximately 2-5 days
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
dollars | 30109 [25077 to 37696] | 27776 [21766 to 37890]

11. Secondary Outcome: Incidence of Adverse Events
Description: Reported as the number participants reporting one or more adverse events on each study arm.
Time Frame: Up to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
Participants | 0 | 1

12. Secondary Outcome: Operating Room Time
Description: Length of time from when the patient entered the operating room to when they left.
Time Frame: Approximately 8 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
hours | 6.2 [4.7 to 7.5] | 5.8 [4.3 to 7.6]

13. Secondary Outcome: Surgical Time
Description: Time from first incision to surgical site closure.
Time Frame: Approximately 8 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
hours | 4.5 [3.3 to 6.0] | 4.4 [2.9 to 5.8]

14. Secondary Outcome: Pain Management
Description: Pharmaceutical costs associated with pain management.
Time Frame: Whole hospitalization, approximately 2-5 days
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
dollars | 830 [692 to 1196] | 807 [630 to 1101]

15. Other Pre Specified Outcome: Quality of Recovery-15 (QoR-15) Total Score
Description: The Quality of Recovery (QoR-15) questionnaire is a 15-item survey that patients rate to measure the quality of their recovery after surgery. Each item in the questionnaire is graded on an 11-point numeric rating scale with total scores ranging from 15 to 150. Higher scores indicate better recovery.
Time Frame: At 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
Number analyzed (Participants) | 59 | 46
score on a scale | 95.5 [77.0 to 105.2] | 104.0 [84.2 to 113.0]

ADVERSE EVENTS:
Time Frame: Up to 24 hours after surgery
Arm/Group | Arm I (Laparotomy, Liposomal Bupivacaine) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/59 | 1/46
Other Adverse Events (participants affected / at risk) | 0/59 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Laparotomy, Liposomal Bupivacaine) (N=59) | Arm II (Laparotomy, Liposomal Bupivacaine, Hydromorphone) (N=46)
Spinal headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT04258631/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT04258631/ICF_001.pdf